CLINICAL TRIAL: NCT06613126
Title: Constructing and Evaluating the Effectiveness of an Intelligent Interaction System for Symptom Management on the Care Needs and Related Factors of Children With Tourette Syndrome and Their Parents
Brief Title: Effectiveness of Symptom Management Application on Parental Care Ability of Children With Tourette Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Mei-Yin Lee, RN PhD Associate professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 202102263B0C601
Record Dates: First submitted 2024-09-22; First posted 2024-09-25 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Tourette Syndrome; Tic Disorder; Neurodevelopmental Disorder
Keywords: symptom management; Application; parent; children with Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders; Neurodevelopmental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- symptom management APP group (Experimental): The experimental group(parents of children with TS between 6 and 12 years old) received TS symptom management APP intervention for four weeks. The experimental group recorded the patterns and treatments of tics at least twice a week and completed relevant readings on TS care information during these four weeks.
  Interventions: Behavioral: Symptom Management APP group
- Health education instructions group (Active Comparator): The control group(parents of children with TS between 6 and 12 years old) continued to receive outpatient verbal and paper health education guidance from healthcare providers.
  Interventions: Other: health education instructions group

INTERVENTIONS:
Behavioral: Symptom Management APP group — Based on symptom management theory and the relevant literature, the researcher designed a symptom management APP. The APP includes a symptom recording system, symptom management skills, and Tourette Syndrome knowledge information to facilitate parents' and children's joint learning.
  Arms: symptom management APP group
Other: health education instructions group — To receive outpatient verbal and paper health education guidance from healthcare providers.
  Arms: Health education instructions group

SUMMARY:
This study developed a Tourette Syndrome (TS) symptom management application (APP) to improve the care needs, sleep quality, anxiety, quality of life, and parenting relationship of parents of children with Tourette Syndrome.

DETAILED DESCRIPTION:
Tourette syndrome (TS) is a common chronic neurodevelopmental disorder in children. Parents play critical roles in helping to manage their child's symptoms, leading to several issues associated with care needs and the parent-child interaction. This study adopted a randomized control study design. The investigators developed a TS symptom management APP based on symptom management theory and the relevant literature. The research subjects were parents of children with TS between 6 and 12 years old. The experimental group received TS symptom management APP intervention for four weeks. The experimental group recorded the patterns and treatments of tics at least twice a week and completed relevant readings on TS care information during these four weeks. The control group continued to receive outpatient verbal and paper health education guidance from healthcare providers. The participants in both groups were requested to complete the following questionnaires, including the care needs scale, WHOQOL-BREF, Pittsburgh Sleep Quality Index (Chinese version), Beck Anxiety Inventory (Chinese version), Parent-Child Relationship Quality Inventory, and the Yale Global Tic Severity Scale. These questionnaires were completed before the intervention and directly after the four-week intervention. The participants were completed again one month and three months after the intervention. To understand the users' satisfaction with this APP, only the participants in the experimental group were requested to complete the Inventory of Technology Acceptance Model when completing the questionnaires during the third posttest. The goal was to strengthen parents' symptom management ability and improve their psychosocial functions and children's disease severity.

ELIGIBILITY:
Inclusion Criteria:

1. Parents of children between 6-12 years old who are diagnosed with Tourette Syndrome by pediatricians.
2. Parents who are the primary caregivers
3. Parents with normal cognitive functioning who can communicate in Mandarin.

Exclusion Criteria:

1. Children with Tourette Syndrome who are suffering from intellectual disability or critical diseases.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Care needs scale for parents of children with Tourette Syndrome (CNS-PCTS) | Change from baseline degree of CNS-PCTS after intervention, 1 month and 3 months.
  The CNS-PCTS contained 13 items, with a score range of 13 to 52. A higher CNS-PCTS score indicated that the parents required greater care needs.
Parent-Child Relationship Quality Inventory | Change from baseline degree of parent-child relationship quality inventory after intervention, 1 month and 3 months.
  The parent-child relationship quality inventory contained 30 items, with a score range of 20 to 100. A higher parent-child relationship quality inventory indicated that the parents perceived greater parent-child relationship quality.

SECONDARY OUTCOMES:
Short version of the World Health Organization Quality of Life (WHOQOL-BREF) | Change from baseline degree of WHOQOL-BREF after intervention, 1 month and 3 months.
  The WHOQOL-BREF contained 28 items, with a score range of 28 to 140. A higher WHOQOL-BREF score indicated that the parents perceived a better quality of life.
Pittsburgh Sleep Quality Index (Chinese version) | Change from baseline degree of Pittsburgh Sleep Quality Index (Chinese version) after intervention, 1 month and 3 months.
  The scoring range is 0-21; a total score above 5 represents poor sleep quality, a score below or equal to 5 means good sleep quality.
Beck Anxiety Inventory (Chinese version) | Change from baseline degree of Beck Anxiety Inventory (Chinese version) after intervention, 1 month and 3 months.
  There are 21 items in the Beck Anxiety Inventory (Chinese version), which measures the severity of anxiety by subjects' self-report.
Yale Global Tic Severity Scale(YGTSS) | Change from baseline degree of YGTSS after intervention, 1 month and 3 months.
  The Yale Global Tic Severity Scale will used in this research to evaluate adolescents' tic severity. The Yale Global Tic Severity Scale has a total score ranging from 0 to 100, with the high score indicating a higher tics severity.

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Yin Lee, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee MY. Living with tics: Nursing care of pediatric tourette syndrome. Biomed J. 2022 Apr;45(2):280-285. doi: 10.1016/j.bj.2021.10.011. Epub 2021 Oct 25. PMID 34710638
- [Result] Lee MY, Wang HS, Chen CJ. Psychosocial experiences in youth with Tourette syndrome: a systematic review and meta-synthesis. Eur Child Adolesc Psychiatry. 2024 Nov;33(11):3787-3802. doi: 10.1007/s00787-023-02339-w. Epub 2023 Dec 21. PMID 38129352
- [Result] Evans GA, Wittkowski A, Butler H, Hedderly T, Bunton P. Parenting Interventions for Children with Tic Disorders: Professionals' Perspectives. J Child Fam Stud. 2016;25:1594-1604. doi: 10.1007/s10826-015-0317-1. Epub 2015 Nov 14. PMID 27110085
- [Result] Ludlow AK, Brown R, Schulz J. A qualitative exploration of the daily experiences and challenges faced by parents and caregivers of children with Tourette's syndrome. J Health Psychol. 2018 Dec;23(14):1790-1799. doi: 10.1177/1359105316669878. Epub 2016 Sep 28. PMID 27682339
- [Result] Pringsheim T, Okun MS, Muller-Vahl K, Martino D, Jankovic J, Cavanna AE, Woods DW, Robinson M, Jarvie E, Roessner V, Oskoui M, Holler-Managan Y, Piacentini J. Practice guideline recommendations summary: Treatment of tics in people with Tourette syndrome and chronic tic disorders. Neurology. 2019 May 7;92(19):896-906. doi: 10.1212/WNL.0000000000007466. PMID 31061208
- [Result] Ricketts EJ, Wolicki SB, Danielson ML, Rozenman M, McGuire JF, Piacentini J, Mink JW, Walkup JT, Woods DW, Bitsko RH. Academic, Interpersonal, Recreational, and Family Impairment in Children with Tourette Syndrome and Attention-Deficit/Hyperactivity Disorder. Child Psychiatry Hum Dev. 2022 Feb;53(1):3-15. doi: 10.1007/s10578-020-01111-4. Epub 2021 Jan 1. PMID 33385257